CLINICAL TRIAL: NCT03490591
Title: The Effects on Hand Function With Robot-assisted Rehabilitation for Children With Cerebral Palsy: a Pilot Study
Brief Title: Robot-assisted Hand Rehabilitation for Children With Cerebral Palsy: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMU-JIRB N201711070
Record Dates: First submitted 2018-02-08; First posted 2018-04-06 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2018-02

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Robotic rehabilitation; Hand function; Activities of Daily Living
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic-assisted intervention (Experimental): In the Robotic-assisted intervention :12 training sessions of Robot-assisted hand rehabilitation(60 minutes a time, 2 times a week)
  Interventions: Behavioral: Robot-assisted hand rehabilitation

INTERVENTIONS:
Behavioral: Robot-assisted hand rehabilitation — Robot-assisted hand rehabilitation: 20 minute of warm-up exercise and 40 minute of robot-assisted hand exercise intervention. Robot-assisted hand exercises include passive range of motion of hand, bilateral hands task, robot-assisted task, and game task.

SUMMARY:
Objective: To investigate the effects of robot-assisted hand rehabilitation with a Gloreha device on hand function and the participation of ADL for children with cerebral palsy(CP).

Materials and Methods: Five children with CP aged 6 to 18 years were recruited and received 12times of robot-assisted hand rehabilitation for 6 weeks of treatment (Sixty minutes a time, twice a week). The performance was assessed by a assessor for three times (pre-test, post-test, follow up at one month). The outcome measures Fugl-Meyer Assessment-Upper Limb section(FMA-UE),Box and block test(BBT), Maximal voluntary contraction(MVC) of extensor digitorum communis(EDC), Flexor digitorum(FD), Grasp strength, & ABILHAND-Kids for ADL ability. Collected data will be analyzed with ANOVA test by SPSS version 20.0, and alpha level was set at .05. Our hypothesis are robot-assisted hand rehabilitation with a Gloreha device has positive effects on hand function and the participation of ADL for children with CP.

DETAILED DESCRIPTION:
Hand function is the most important for ADL and learning ability. Many cerebral palsy(CP) suffered problems with the gross motor dysfunction and hand function disability. An inability to use the upper extremity in daily life can lead to loss of independence with ADLs and of important occupations (eg, school). Robotic therapy can deliver larger amounts of upper extremity movement practice for these individuals. Although the Robotic therapy appears to provide some benefit for upper extremity motor abilities and participation but is of uncertain utility for cerebral palsy(CP).

Objective: To investigate the effects of robot-assisted hand rehabilitation with a Gloreha device on hand function and the participation of ADL for children with cerebral palsy(CP).

Five children with CP aged 6 to 18 years were recruited and received 12times of robot-assisted hand rehabilitation for 6 weeks of treatment (Sixty minutes a time, twice a week). The performance was assessed by a assessor for three times (pre-test, post-test, follow up at one month). The outcome measures Fugl-Meyer Assessment-Upper Limb section(FMA-UE),Box and block test(BBT), Maximal voluntary contraction(MVC) of extensor digitorum communis(EDC), Flexor digitorum(FD), grasp strength, & ABILHAND-Kids for ADL ability. Collected data will be analyzed with ANOVA test by SPSS version 20.0, and alpha level was set at .05. Our hypothesis are robot-assisted hand rehabilitation with a Gloreha device has positive effects on hand function and the participation of ADL for children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy(CP) or stroke
* Age younger than 18 and older than 6 years old
* Could follow 2 step order instruction
* No Botulinum injection during the recent 6 month and the experiment period
* Chronicity > 1 years and stable medicine condition
* Could sit steady after the position

Exclusion Criteria:

* Individuals with other medical symptoms that can affect movement
* Individuals with visual or auditory impairment who couldn't see or hear the feedback from the device clearly

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment:Upper Limb section | Change from baseline to 6 weeks, follow up at one month
  The Fugl-Meyer motor assessments for the upper limb section(scores from 0 to 66 points)that evaluates reflexes, volitional movements and rapid alternating movements. The higher values represent a better outcome.

SECONDARY OUTCOMES:
Box and block test | Change from baseline to 6 weeks, follow up at one month
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. Clients are scored based on the number of blocks transferred from one compartment to the other compartment in 60 seconds. Score each hand separately. Higher scores are indicative of better manual dexterity.
EMG: record maximal voluntary contraction(MVC) of brachioradialis, extensor carpi | Change from baseline to 6 weeks, follow up at one month
  Surface electromyography root mean square from brachioradialis and extensor carpi was normalized to the maximal voluntary contraction recording. The higher muscle activation during the task indicate the more efficacy to grasp or release the block.
Jamar Handgrip Dynamometer | Change from baseline to 6 weeks, follow up at one month
  The Jamar hydraulic handgrip dynamometer for measuring the maximum isometric strength of the hand and forearm muscles. The mean score among three trials of each instrument was recorded for data calculations. The higher scores presents the better hand grip strength.
ABILHAND-Kids questionnaire | Change from baseline to 6 weeks, follow up at one month
  A measure of manual ability for children with upper limb impairments. The scale measures a person's ability to manage daily activities that require the use of the upper limbs, whatever the strategies involved. The parent is asked to rate his/her perception on the response scale as "Impossible", "Difficult" or "Easy" (0 = "Impossible", 1 = "Difficult" or 2 = "Easy"). The activities not attempted by the child within the last 3 months are not scored and are entered as not applicable. The total score based on 21 activities is then converted into a linear measure of manual ability (logits). This test was specifically developed for children with CP using the Rasch measurement model and showed a good reliability and reproducibility over time.

CONTACTS AND LOCATIONS:
Overall Officials: Jui chi Lin, master, Study Chair — Taipei Medical University, Taiwan, R.O.C.
Locations (1):
- Department of Physical Medicine and Rehabilitation, Shuang Ho Hospital, Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bax M, Goldstein M, Rosenbaum P, Leviton A, Paneth N, Dan B, Jacobsson B, Damiano D; Executive Committee for the Definition of Cerebral Palsy. Proposed definition and classification of cerebral palsy, April 2005. Dev Med Child Neurol. 2005 Aug;47(8):571-6. doi: 10.1017/s001216220500112x. PMID 16108461
- [Background] Novak I. Evidence-based diagnosis, health care, and rehabilitation for children with cerebral palsy. J Child Neurol. 2014 Aug;29(8):1141-56. doi: 10.1177/0883073814535503. Epub 2014 Jun 22. PMID 24958005
- [Background] Arner M, Eliasson AC, Nicklasson S, Sommerstein K, Hagglund G. Hand function in cerebral palsy. Report of 367 children in a population-based longitudinal health care program. J Hand Surg Am. 2008 Oct;33(8):1337-47. doi: 10.1016/j.jhsa.2008.02.032. PMID 18929198
- [Background] Sakzewski L, Ziviani J, Boyd RN. Efficacy of upper limb therapies for unilateral cerebral palsy: a meta-analysis. Pediatrics. 2014 Jan;133(1):e175-204. doi: 10.1542/peds.2013-0675. Epub 2013 Dec 23. PMID 24366991
- [Background] Varalta V, Picelli A, Fonte C, Montemezzi G, La Marchina E, Smania N. Effects of contralesional robot-assisted hand training in patients with unilateral spatial neglect following stroke: a case series study. J Neuroeng Rehabil. 2014 Dec 5;11:160. doi: 10.1186/1743-0003-11-160. PMID 25476507
- [Background] Sgaggio, E., Joint and functional benefits of a robotic glove for post-stroke patients. publication pending, 2015
- [Background] Fasoli SE, Fragala-Pinkham M, Hughes R, Hogan N, Krebs HI, Stein J. Upper limb robotic therapy for children with hemiplegia. Am J Phys Med Rehabil. 2008 Nov;87(11):929-36. doi: 10.1097/PHM.0b013e31818a6aa4. PMID 18936558
- [Background] Ming-Juei Chang (2017).Prevalence, healthcare and rehabilitation services utilization in individuals with cerebral palsy.Taiwan Master Master's Thesis
- [Background] Levitt, S. (2013). Treatment of cerebral palsy and motor delay. John Wiley & Sons.
- [Background] Ching-Yi Chen,Ching-Chun Li,Jiunn-Horng Kang(2013). Medical Utilization among Patients with Cerebral Palsy, Taiwan Journal of Physical Medicine and Rehabilitation41(4), 225-234.
- [Background] McHale K, Cermak SA. Fine motor activities in elementary school: preliminary findings and provisional implications for children with fine motor problems. Am J Occup Ther. 1992 Oct;46(10):898-903. doi: 10.5014/ajot.46.10.898. PMID 1463061
- [Background] Asher AV. Handwriting instruction in elementary schools. Am J Occup Ther. 2006 Jul-Aug;60(4):461-71. doi: 10.5014/ajot.60.4.461. PMID 16915877
- [Background] Henderson, A., & Pehoski, C. (Eds.). (2006). Hand function in the child: Foundations for remediation. Elsevier Health Sciences.
- [Background] Hsieh-Chun Hsieh(2010). Effects of Parent-Child Toy-Playing Activities on the Motor Development of Children with Cerebral Palsy. Ulletin of special education, 35(2), 81-101.
- [Background] Huang, C. W. (2016). Effectiveness of unilateral versus bilateral intensive training in children with cerebral palsy: a randomized controlled study. Taiwan University Occupational Therapy Research Institute Thesis, 1-82.
- [Background] Lohse KR, Hilderman CG, Cheung KL, Tatla S, Van der Loos HF. Virtual reality therapy for adults post-stroke: a systematic review and meta-analysis exploring virtual environments and commercial games in therapy. PLoS One. 2014 Mar 28;9(3):e93318. doi: 10.1371/journal.pone.0093318. eCollection 2014. PMID 24681826
- [Background] Lohse K, Shirzad N, Verster A, Hodges N, Van der Loos HF. Video games and rehabilitation: using design principles to enhance engagement in physical therapy. J Neurol Phys Ther. 2013 Dec;37(4):166-75. doi: 10.1097/NPT.0000000000000017. PMID 24232363
- [Background] Pichierri G, Wolf P, Murer K, de Bruin ED. Cognitive and cognitive-motor interventions affecting physical functioning: a systematic review. BMC Geriatr. 2011 Jun 8;11:29. doi: 10.1186/1471-2318-11-29. PMID 21651800
- [Background] Winkels DG, Kottink AI, Temmink RA, Nijlant JM, Buurke JH. Wii-habilitation of upper extremity function in children with cerebral palsy. An explorative study. Dev Neurorehabil. 2013;16(1):44-51. doi: 10.3109/17518423.2012.713401. Epub 2012 Oct 3. PMID 23030054
- [Background] Acar G, Altun GP, Yurdalan S, Polat MG. Efficacy of neurodevelopmental treatment combined with the Nintendo((R)) Wii in patients with cerebral palsy. J Phys Ther Sci. 2016 Mar;28(3):774-80. doi: 10.1589/jpts.28.774. Epub 2016 Mar 31. PMID 27134357
- [Background] Dobkin BH. Strategies for stroke rehabilitation. Lancet Neurol. 2004 Sep;3(9):528-36. doi: 10.1016/S1474-4422(04)00851-8. PMID 15324721
- [Background] Buerger, S. P., & Hogan, N. (2006, October). Relaxing passivity for human-robot interaction. In Intelligent Robots and Systems, 2006 IEEE/RSJ International Conference on (pp. 4570-4575). IEEE.
- [Background] Volpe BT, Lynch D, Rykman-Berland A, Ferraro M, Galgano M, Hogan N, Krebs HI. Intensive sensorimotor arm training mediated by therapist or robot improves hemiparesis in patients with chronic stroke. Neurorehabil Neural Repair. 2008 May-Jun;22(3):305-10. doi: 10.1177/1545968307311102. Epub 2008 Jan 9. PMID 18184932
- [Background] Pětioký, J. Robot-assisted therapy integrated with virtual reality for rehabilitation of hand function after stroke: a clinical case study. in the 20th ESPRM Congress 2016.
- [Background] Vanoglio F, Bernocchi P, Mule C, Garofali F, Mora C, Taveggia G, Scalvini S, Luisa A. Feasibility and efficacy of a robotic device for hand rehabilitation in hemiplegic stroke patients: a randomized pilot controlled study. Clin Rehabil. 2017 Mar;31(3):351-360. doi: 10.1177/0269215516642606. Epub 2016 Jul 10. PMID 27056250
- [Background] Lincoln, N. B., Jackson, J. M., & Adams, S. A. (1998). Reliability and revision of the Nottingham Sensory Assessment for stroke patients. Physiotherapy, 84(8), 358-365.